CLINICAL TRIAL: NCT04718064
Title: Revascularization Pretreated With Fingolimod in Acute Stroke
Acronym: REPAIR FAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XYFY00001
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fingolimod with standard therapy (Experimental): Patients will be treated with intravascular therapy and fingomod.
  Interventions: Drug: Fingolimod
- Placebo with standard therapy (Placebo Comparator): Patients will be treated with intravascular therapy and placebo.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Fingolimod — fingolimod (Gilenya, Novartis) at a dosage of 0.5 mg once daily, for three consecutive days
  Arms: fingolimod with standard therapy
Drug: placebo — placebo once daily, for three consecutive days,
  Arms: Placebo with standard therapy

SUMMARY:
Acute ischemic stroke (AIS) is a common type of stroke in the elderly. Timely blood flow recovery can effectively improve the long-term prognosis of patients. According to five large-scale multicenter randomized controlled trials (MR clean, swift-prime, revascat, escape and extend-ia) in recent years, the effect of endovascular therapy (EVT) for acute anterior circulation occlusion of great vessels is significantly better than that of drug therapy alone. Therefore, for patients who meet the "Chinese guidelines for the diagnosis and treatment of acute ischemic stroke" (2018 Edition), the effect of EVT is better than that of drug therapy alone, Intravenous thrombolysis within 4.5 hours and endovascular mechanical thrombectomy within 6 hours can effectively relieve the clinical symptoms and reduce the mortality of AIS. However, due to the narrow application time window of intravenous thrombolysis and mechanical thrombectomy, although the thrombectomy time window of some eligible patients was relaxed to 24 hours after dawn and defuse3 and other related studies, the reperfusion injury after the blocked cerebral artery recanalization has brought huge obstacles to clinical application. Therefore, how to improve the prognosis of patients with endovascular therapy has become a hot research direction.

Fingomod is a kind of sphingosine analogues acting on sphingosine-1-phosphate (sipr). After phosphorylation in the body, fingomod combines with lymphocyte SIP receptor, changes lymphocyte migration route, prevents it from entering the area outside the lymphoid tissue, so as to avoid its infiltration into the central nervous system and achieve immunosuppression. Currently, it is the first-line disease modifying oral drug for multiple sclerosis. Fingolmod shows neuroprotective effects on many central nervous system diseases including cerebral ischemia. Fingomod not only reduced the number of lymphocytes invading the brain, but also decreased the number of lymphocytes in the microcirculation system

ELIGIBILITY:
Inclusion Criteria:

* The patient was over 18 years old;
* The NIHSS score was < 30 and NIHSS > 5;
* CTA / MRA / DSA confirmed occlusion of M1 segment of internal carotid artery or middle cerebral artery, and aspect score ≥ 6;
* CTP or MRI showed mismatch (ischemic core volume < 70ml, CTP mismatch > 1.2
* Normal to random time within 24 hours
* Written informed consent signed by patients or their families

Exclusion Criteria:

* Standard contraindications to alteplase or mechanical thrombectomy
* Cerebral hemorrhage confirmed by imaging
* Cardiovascular diseases (such as bradycardia, etc.)
* Systolic blood pressure > 185mmhg or diastolic blood pressure > 110mmhg, and oral antihypertensive drugs can not be controlled
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
90 day mRS score | at day 90
  recovery

SECONDARY OUTCOMES:
mRS score of 0-1 (%) | at day 90
  excellent recovery
mRS score of 1-2 (%) | at day 90
  general recovery
Recanalization success rate | from baseline to 2 day
  baseline mTICI score - 2 day mTICIS score
the growth in infarct volume (mL) | from 24 hour to 7 day
  24 hour DWI infarct volume (mL) - 7 day FLAIR infarct volume (mL)
the penumbral salvage volume (mL) | from baseline to 1 day
  baseline CTP hypoperfusion volume (mL) - 24 hour DWI infarct volume (mL)
the change on the NIHSS score | from baseline to 1 day
  baseline NIHSS score - 1 day NIHSS score
the change on the NIHSS score | from baseline to 7 day
  baseline NIHSS score - 7 day NIHSS score baseline NIHSS score - 7 day NIHSS score baseline NIHSS score - 7 day NIHSS score
the change on the EQ-5D score | from baseline to 90 day
  baseline EQ-5D score - 90 day EQ-5D score

IPD SHARING:
Plan to Share IPD: No